CLINICAL TRIAL: NCT02881203
Title: BRAVEHeart - Breast Radiotherapy Audio Visual Enhancement for Sparing the Heart
Brief Title: Breast Radiotherapy Audio Visual Enhancement for Sparing the Heart
Acronym: BRAVEHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAVEHeartV1
Record Dates: First submitted 2016-08-22; First posted 2016-08-26 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; radiation; DIBH; cardiac toxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathe Well + RPM (Experimental): Participants will receive Breathe Well audiovisual feedback in addition to the RPM system
  Interventions: Device: Breathe Well; Device: RPM
- RPM (Active Comparator): Varian's RPM system is the current standard of care at Royal North Shore Hospital where this trial is to be run.
  Interventions: Device: RPM

INTERVENTIONS:
Device: Breathe Well — Breathe Well is an audiovisual biofeedback device used to assist patients to regulate their breathing whilst undergoing radiation treatment.
  Arms: Breathe Well + RPM
Device: RPM — Varian Real-time Position Management (RPM) system

SUMMARY:
This study investigates the Breathe Well device to test whether it is superior to the existing treatment standard of the Varian Realtime Position Management (RPM) system in assisting patients with deep inspiration breath hold.

DETAILED DESCRIPTION:
Recent studies have demonstrated an increased risks of cardiac disease in breast cancer radiotherapy patients. For patients diagnosed <50 years old, the risks for cardiovascular diseases/events were increased by 24-82% comparing left and right breast radiotherapy. The deep inspiration breath hold (DIBH) technique addresses this problem by reducing the heart dose by up to half, thus potentially reducing the increased rate of major coronary events by 20%. Providing patients with visual feedback in addition to audio guidance has been demonstrated to improve the reproducibility of the DIBH technique by 95% and stability by 80%.

Breathe Well is a new audiovisual feedback device that may increase the accuracy and workflow of implementing DIBH for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Left-sided breast cancer patients (invasive and in situ)
* Supine positioning of the patients.
* Ability to perform a ≥20s breath hold
* >18 years old
* An ECOG score in the range of 0 to 2
* Able to give written informed consent and willingness to participate and comply with the study
* Patients must be able to read and complete questionnaires in English

Exclusion Criteria:

* Involvement or at risk regional lymph nodes
* Pregnant / lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of Breathe Well | 2 years
  The accuracy will be measured by comparing 'Breathe Well' and RPM measurements with images acquired of the breast during the radiation treatment using an electronic portal imaging device (EPID).

SECONDARY OUTCOMES:
Difference in set up times for Breathe Well vs RPM | 2 years
  The setup times for both systems, the 'Breathe Well' and the modified RPM system; will be measured for all fractions.
Patient comfort | 2 years
  To investigate patient comfort in using 'Breathe Well' via a patient survey.
Staff perception of Breathe Well | 2 years
  To investigate staff perception of 'Breathe Well' via a technology assessment survey.
To develop the use of EPID for real time MLC tracking during breast radiotherapy | 2 years
To compare actual and planned doses | 2 years
  Using dose reconstruction estimate the dose distribution delivered during radiotherapy and compare this with the planned dose.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Lamoury, Medicine, Principal Investigator — Royal North Shore Hospital
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available to researchers upon request, once evidence of ethical approval has been provided.

REFERENCES:
- [Derived] Byrne HL, Steiner E, Booth J, Lamoury G, Morgia M, Richardson K, Ambrose L, Makhija K, Stanton C, Zwan B, Bromley R, Atyeo J, Silvester S, Plant N, Keall P. BRAVEHeart: a randomised trial comparing the accuracy of Breathe Well and RPM for deep inspiration breath hold breast cancer radiotherapy. Trials. 2023 Feb 22;24(1):132. doi: 10.1186/s13063-023-07072-y. PMID 36814310